CLINICAL TRIAL: NCT04444817
Title: Evaluation of the Impact of Tacrolimus-based Immunosuppression on Heidelberg Liver Transplant Cohort (HDTACRO): Study Protocol for an Investigator Initiated, Non-interventional Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. A. Mehrabi, Professsor, Head of the Division of Liver Surgery and Visceral Transplantation, University Hospital Heidelberg
Other Study IDs: S-260/2018
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Liver Transplantation
Keywords: Tacrolimus; immunosuppression; Liver transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tacrolimus-based immunosuppression: Similar to the clinical routine, as soon as a patient is able to swallow and has a sufficient gastrointestinal activity, Tacrolimus-based immunosuppression using Prograf®, Advagraf® or Envarsus® will be started.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Similar to the clinical routine, as soon as a patient is able to swallow and has a sufficient gastrointestinal activity, Tacrolimus-based immunosuppression using Prograf®, Advagraf® or Envarsus® will be started. Furthermore, calcineurin inhibitors-based immunosuppression will be used (initial dose based on the patients' body weight) with the goal of tough levels of 3-7 ng/mL in the first seven days after liver transplantion, depending on immune status and indication for transplantation. Further tough levels will be determined based on factors such as patients' history and indication for liver transplant.

SUMMARY:
Modern immunosuppression is characterized by a combination of different immunosuppressants. As a result, the dose of the individual substances, and thus also their side effects can be reduced. Immunosuppression on the basis of low-dose calcineurin inhibitors (CNI) with comparatively low CNI target levels could therefore prevail. Despite all efforts to optimize the treatment regimen after liver transplantation from deceased donors, the amount of medication remains high throughout the postoperative course with CNIs being the main component of immunosuppressive treatment. The main substance used is Tacrolimus in combination with steroids and possibly Mycophenolic acid. Tacrolimus is considered a narrow therapeutic index drug requiring individual dose titration, to achieve a satisfactory balance between maximizing efficacy and minimizing dose-related toxicity. Furthermore, transplanted recipients have to remain to a very demanding medication regimen for a long time. The burden of pills required is associated with decreased adherence, and lack of adherence can lead to rejection and possibly graft loss. The aim of present study is to assess the tough levels and need of doses adaptation in de novo liver transplantation with Tacrolimus in the clinical routine, without any intervention in the treatment regimen.

DETAILED DESCRIPTION:
Tacrolimus is considered a narrow therapeutic index drug requiring individual dose titration, to achieve a satisfactory balance between maximizing efficacy and minimizing dose-related toxicity. The pharmacokinetic profile of Tacrolimus is characterized by a high degree of inter- and intraindividual variability. Although it is rapidly absorbed, the bioavailability of Tacrolimus in the twice-daily capsule formulation is low and variable, ranging from 17 to 23%. This could be due to poor water solubility, extensive first pass metabolism, p-glycoprotein-mediated efflux and the ingestion of food. Tacrolimus twice-daily capsules are also associated with a characteristic high peak following dosing, which may be associated with increased toxicity.

Furthermore, transplanted recipients have to remain to a very demanding medication regimen for a long time. The burden of pills required is associated with decreased adherence, and lack of adherence can lead to rejection and possibly graft loss.

The development of once-daily Tacrolimus forms without any change of the form of dissolving has already been shown to increase patients' adherence, while little difference has been demonstrated in the Tacrolimus pharmacokinetic profile. The pharmacokinetic profile of Tacrolimus is characterized by flatter kinetics (i.e., less fluctuation and swing) compared to twice-daily Tacrolimus providing for a balanced concentration-time consistency over 24 hours which can also lead to reduced incidence and/or intensity of drug toxicity-related adverse events. Since the development of LCP-Tacrolimus once-daily tablets, with the use of MeltDose® technology, clinical data have shown lower peak and reduced peak-to-tough fluctuations.

ELIGIBILITY:
Inclusion Criteria:

* 18 < Recipient Age ≤ 60 years old
* Ability to understand and sign an informed consent form
* Operation and immediate post-operative therapy within the Department of General, Visceral and Transplantion Surgery, University Hospital Heidelberg
* De novo liver transplantation until POD 7
* Immunosuppression after liver transplantation based on Tacrolimus

Exclusion Criteria:

* Re-transplantation
* Acute infection of the biliary tract, pneumonia or CMV infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: One hundred Recipients who underwent de novo liver transplant and treated with various oral Tacrolimus-based immunosupresions (Prograf®, Advagraf® and Envarsus®)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of required dose adjustments of Tacrolimus formulations used in clinical routine for achieving the target tough level | Six months

SECONDARY OUTCOMES:
Tacrolimus tough level | Six months
Tacrolimus dosing | Six months
Concentration/dose ratio | Six months
Mean cumulative dose for cost analysis | Six months
Routine laboratory tests | Six months
Survival rate | Six months
The incidence of acute rejection | Six months
The incidence of re-transplantation | Six months
Patients' therapy adherence | Six months
The incidence of infection with need to reduce Immunosuppression | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Visceral Transplantation, Department of General, Visceral andTransplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khajeh E, Polychronidis G, Ramouz A, Alamdari P, Lemekhova A, Saracevic M, Ali-Hasan-Al-Saegh S, Ghamarnejad O, Majlesara A, Abbasi Dezfouli S, Nickkholgh A, Weiss KH, Rupp C, Mehrabi A, Mieth M. Evaluation of the impact of Tacrolimus-based immunosuppression on Heidelberg liver transplant cohort (HDTACRO): Study protocol for an investigator initiated, non-interventional prospective study. Medicine (Baltimore). 2020 Sep 25;99(39):e22180. doi: 10.1097/MD.0000000000022180. PMID 32991411